CLINICAL TRIAL: NCT01006486
Title: Evaluation of Impact of the Implantation of an Anticoagulation Clinic in an University Hospital in Brazil
Brief Title: Outcomes of an Anticoagulation Clinic in an University Hospital
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Professor Antonio Luiz Pinho Ribeiro, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: COEP376/09
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Cardiopathy; Chagas Disease; Hemorrhage; Thrombosis
Keywords: Oral anticoagulants; Warfarin; Anticoagulation clinic; Thrombosis; Hemorrhage
MeSH Terms: conditions — Heart Diseases; Chagas Disease; Hemorrhage; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anticoagulation clinic (Experimental): Anticoagulation clinic, including all procedures related to a standardized use of coumarins.
  Interventions: Other: Anticoagulation clinic
- Standard care (Active Comparator): Standard use of coumarins, as prescribed by their physicians.
  Interventions: Other: Standard anticoagulation care

INTERVENTIONS:
Other: Anticoagulation clinic — Patients randomized to this arm will be cared at an anticoagulation clinic, with educational measures and standardized procedures related to the use of coumarins.
  Other Names: Implementation of a health service
  Arms: Anticoagulation clinic
Other: Standard anticoagulation care — Patients randomized to this arm will be cared by their physician, with standard care. No standardized protocol of the use of coumarins will be established.
  Other Names: Implementation of a health service
  Arms: Standard care

SUMMARY:
A clinical trial designed to compare the oral anticoagulation control obtained by an anticoagulation clinic and the usual medical care in Chagas and Non-Chagas disease patients.

DETAILED DESCRIPTION:
A Randomized, Crossover, Clinical Trial performed to compare the results of oral anticoagulation for Chagas and non-Chagas disease patients treated at an anticoagulation clinic and by the usual clinical practice. The primary endpoint was the time that the International Normalized Ratio (INR) was in the therapeutic range and the secondary endpoints were thromboembolic/haemorragic events.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Chagas and non-Chagas disease patients
* Any indication for chronic treatment with warfarin
* Anticoagulation for at least 30 days.

Exclusion Criteria:

* Refusal to participate in the study;
* Use of phenprocoumon;
* Expectation of treatment lower than 1 year;
* Difficulties to attend medical visits;
* Participation in other prospective clinical study involving anticoagulation care during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range | 1 year

SECONDARY OUTCOMES:
Hemorrhagic events | 1 year
Thromboembolic events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio L Ribeiro, MD, PhD, Study Chair — Federal University of Minas Gerais; Manoel Otávio C Rocha, MD, PhD, Principal Investigator — Federal University of Minas Gerais; Maria Auxiliadora P Martins, Pharmacist, Principal Investigator — Federal University of Minas Gerais; Cibele C César, MD, PhD, Principal Investigator — Federal University of Minas Gerais; Daniel D Ribeiro, Physician, Principal Investigator — Federal University of Minas Gerais; Vandack Nobre, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil